CLINICAL TRIAL: NCT03143465
Title: MR-Angiografi (MRA) og MR-Spektroskopi (MRS) Hos Raske forsøgspersoner og Patienter Med migræne Uden Aura Provokeret Med Calcitonin Gen-relateret Peptid (CGRP) og Sildenafil
Brief Title: Pharmacologically Triggered Migraine Without Aura and Neuroimaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Samaira Younis, MD, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-15019063
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Migraine With Aura
MeSH Terms: conditions — Migraine with Aura | interventions — Calcitonin Gene-Related Peptide; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No

ARMS (3):
- CGRP (Experimental)
  Interventions: Drug: Calcitonin Gene-Related Peptide
- Sildenafil (Experimental)
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitonin Gene-Related Peptide
  Arms: CGRP
Drug: Sildenafil
  Arms: Sildenafil
Drug: Placebo
  Arms: Placebo

SUMMARY:
Migraine is a highly disabling disorder affecting 14% of the general population Worldwide and ranked as the 6th most debilitating disease worldwide by the WHO. One of the most fundamental questions of migraine, which remains to be elucidated, is the mechanism behind the generation of migraine attacks.

The investigators will use calcitonin gene-related peptide (CGRP) and sildenafil as pharmacological triggers of migraine, combined with advanced neuroimaging techniques, to investigate the attack initiating pathophysiology.

Both substances have previously been administered to healthy participants and migraine without aura patients, inducing headache and migraine-like-attacks.

The investigators hope to contribute with novelty to the current understanding of the migraine pathophysiology and development of more efficient treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* Weight: 50-100 kg
* Diagnosis of migraine without aura (patient group only)
* Attacks of migraine without aura at least once every second month (patient group only)

Exclusion Criteria:

* Inconsistent laterality of headache
* History or family history of migraine (healthy subject group only)
* Tension-type headache more than one day per month on average (healthy subject group only)
* Tension-type headache to such a degree that the episodic migraine diagnosis is no longer fulfilled
* Any other primary headache disorder
* Daily intake of medication (apart from oral contraceptives)
* Intake of any medication less than 4 half-lives before study start
* Daily smoking
* Pregnant or breastfeeding women
* Headache 48 h prior to study day
* Hypertension on the study day (systolic BP>150 mmHg or diastolic BP> 100 mmHg)
* Hypotension on the study day (systolic BP<90 mmHg or diastolic BP<50 mmHg)
* History of any cardiovascular disease including cerebrovascular disease
* Any disorder, that is deemed ineligible for participation by the study physicians
* Contraindications of MRI
* No use of safe contraception (women of fertile age only)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
CGRP and sildenafil induced headache and MRI changes | 0- 12h
  CGRP and sildenafil induced headache and MRI changes

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, University Hospital, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Younis S, Christensen CE, Toft NM, Soborg T, Amin FM, Hougaard A, Ashina M. Investigation of distinct molecular pathways in migraine induction using calcitonin gene-related peptide and sildenafil. Cephalalgia. 2019 Dec;39(14):1776-1788. doi: 10.1177/0333102419882474. Epub 2019 Nov 4. PMID 31684759
- [Derived] Christensen CE, Younis S, Lindberg U, Boer VO, de Koning P, Petersen ET, Paulson OB, Larsson HBW, Amin FM, Ashina M. Ultra-high field MR angiography in human migraine models: a 3.0 T/7.0 T comparison study. J Headache Pain. 2019 May 6;20(1):48. doi: 10.1186/s10194-019-0996-x. PMID 31060491